CLINICAL TRIAL: NCT06998303
Title: Imaging Core Aim 2, and Udall Project 2 Aim 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Udall 2
Record Dates: First submitted 2025-04-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a single arm study in which all participants will receive the same study interventions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): 2 Study Procedures: Patients who have been already implanted with a MRI compatible DBS device (Medtronic Percept / Percept RC™)
  Interventions: Other: Bipolar DBS stimulation

INTERVENTIONS:
Other: Bipolar DBS stimulation — All participants will receive bipolar DBS through stimulation contacts 3 (most dorsal GP contact) and contact 2 (adjacent to contact 3) as specified by the device manufacturer. Bipolar stimulation through contacts 3 and 2 may be different from the settings used by the participant for optimal clinical improvement, as determined by their DBS care provider

SUMMARY:
More than one million people in the United States have Parkinson's disease (PD) and the prevalence is expected to double by 2040. Over 60% of these individuals will develop debilitating postural instability and gait disturbances (PIGD), including freezing of gait (FOG). With disease progression, axial motor symptoms typically become resistant to dopamine replacement therapies (e.g. levodopa) and a primary source of disability and morbidity. While subthalamic (STN) and globus pallidus internus (GPi) deep brain stimulation (DBS) using standard locations and stimulation parameters can be highly effective for the treatment of the cardinalmotorsymptomsof PD, both treatments often fail to control levodopa-resistant motor features of PD such as PIGD. DBS can also impair cognitive function which further exacerbates PIGD, particularly when the task requires attentional resources. Thus, despite considerable improvements in appendicular bradykinesia, rigidity and tremor with conventional DBS, the disease can continue to be dominated by PIGD, leading to increased falls, decreased mobility, and increased rate of hospitalization and morbidity. This is why one of the top NINDS priorities for clinical research in PD is the development of novel therapeutic approaches, such as DBS targeting, to treat levodopa-resistant motor symptoms.

This study will provide crucial information to elucidate the functional properties of the networks involved in Deep Brain Stimulation (DBS) treatment. By refining our understanding of the neural networks involved in stimulation of DBS targets, we will improve our ability to program patients to enhance their clinical outcomes and minimize side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and up
* Implanted with MR-compatible DBS device (Medtronic Percept/Percept RC DBS System) for treatment of Parkinson's disease
* English speaking

Exclusion Criteria:

* Unable to consent for themselves
* Implanted with a DBS device that is not MR compatible
* Pregnant
* Extreme claustrophobia
* Any contraindications for MRI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Oxygen-Level Dependent (BOLD) signal in leg region of primary motor cortex | 8 hours
  Data will be obtained from functional MRI scanning with the participant at rest, with DBS cycling between ON and OFF stimulation.
  The change in BOLD signal in the leg region of the primary motor cortex will be obtained by contrasting signals obtained during ON vs. OFF stimulation states.
  The change in BOLD signal represents the increase/decrease in brain activity in the leg region related to stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Harel, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States